CLINICAL TRIAL: NCT04822233
Title: A Comparative Study of Hall Technique, Modified Hall Technique and Conventional Stainless-Steel Crown Restorations in the Treatment of Primary Molars With Proximal Caries Lesions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nat Salako BDS(Hons), Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-DB-20-1247
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Dental Caries
Keywords: molars
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Hall Technique (HT) (Experimental)
  Interventions: Device: Hall Technique (HT)
- Modified Hall Technique (MHT) (Experimental)
  Interventions: Device: Modified Hall Technique (MHT)
- Conventional Technique (CT) (Active Comparator)
  Interventions: Device: Conventional Technique (CT)

INTERVENTIONS:
Device: Hall Technique (HT) — Prior to each restoration, a bacterial sample of the lesion will be obtained with a cotton swap and dispensed in a transport medium for microbial analyses.The preformed metal crown (PMC) will placed without local anesthetic and without crimping or trimming. When the contact points are tight, an orthodontic elastic separator will be placed for 2 hours prior to PMC placement. The PMCs will be cemented with glass ionomer Ketac cem.
  Arms: Hall Technique (HT)
Device: Modified Hall Technique (MHT) — Prior to each restoration, a bacterial sample of the lesion will be obtained with a cotton swab and dispensed in a transport medium for microbial analyses.This group will in addition to all the procedures for the Hall will have the Caries lesions treated with 30% Silver Diamine Fluoride (SDF) before cementation of the stainless-steel crowns.
  Arms: Modified Hall Technique (MHT)
Device: Conventional Technique (CT) — Prior to each restoration, a bacterial sample of the lesion will be obtained with a cotton swab and dispensed in a transport medium for microbial analyses. Conventional occlusal, proximal slicing and when necessary buccal and lingual surfaces will be carried out under local anesthesia and dental dam isolation local anesthesia.The PMC will be trimmed and crimped at the gingival margin to improve the fit, and cemented with Ketac cem.
  Arms: Conventional Technique (CT)

SUMMARY:
The purpose of this study is to compare the effectiveness of the Hall technique and modified Hall technique to the conventional Stainless-Steel Crown restoration in the treatment of primary molars with dentinal caries with or without proximal ridge intact.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit children
* Children who exhibit cooperative behavior at initial bitewing radiograph procedure
* Children with symptom-free or reversible pulpitis restorable first and second primary molars in both arches
* Teeth with D1 lesions will be included
* No periapical or furcation pathologies on bite wing radiographs

Exclusion Criteria:

* Medically compromised children
* Children with uncooperative behavior during bitewing radiograph process
* Primary molars with irreversible pulpitis
* Teeth with furcation or peri radicular pathologies

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 132 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Success as assessed by number of participants with no coronal or peri-radicular pathology | 3 months post intervention
Success as assessed by number of participants with no coronal or peri-radicular pathology | 6 months post intervention
Success as assessed by number of participants with no coronal or peri-radicular pathology | 9 months post intervention
Success as assessed by number of participants with no coronal or peri-radicular pathology | 12 months post intervention
Amount of time taken to complete the intervention | from start of intervention to end of intervention (about 45 minutes to 11/2 hours)

SECONDARY OUTCOMES:
Number of participants with occlusal contact of the molars as assessed by the strip test | 3 months post intervention
  Measured by passing a strip between the contra-lateral upper and lower posterior natural teeth with the child biting into maximum intercuspation. If the strip passes without resistance between teeth anterior or posterior to the SSC there is no occlusal contact.
Number of participants occlusal contact of the molars as assessed by the strip test | 6 months post intervention
  Measured by passing a strip between the contra-lateral upper and lower posterior natural teeth with the child biting into maximum intercuspation. If the strip passes without resistance between teeth anterior or posterior to the SSC there is no occlusal contact.
Number of participants occlusal contact of the molars as assessed by the strip test | 9 months post intervention
  Measured by passing a strip between the contra-lateral upper and lower posterior natural teeth with the child biting into maximum intercuspation. If the strip passes without resistance between teeth anterior or posterior to the SSC there is no occlusal contact.
Number of participants occlusal contact of the molars as assessed by the strip test | 12 months post intervention
  Measured by passing a strip between the contra-lateral upper and lower posterior natural teeth with the child biting into maximum intercuspation. If the strip passes without resistance between teeth anterior or posterior to the SSC there is no occlusal contact.
Molar height in occlusion | 3 months post intervention
Molar height in occlusion | 6 months post intervention
Molar height in occlusion | 9 months post intervention
Molar height in occlusion | 12 months post intervention
Anterior occlusal contact | 3 months post intervention
  Over lap of the upper and lower incisors will be measured in millimeters.If incisors are missing, canines will be used.
Anterior occlusal contact | 6 months post intervention
  Over lap of the upper and lower incisors will be measured in millimeters.If incisors are missing, canines will be used.
Anterior occlusal contact | 9 months post intervention
  Over lap of the upper and lower incisors will be measured in millimeters.If incisors are missing, canines will be used.
Anterior occlusal contact | 12 months post intervention
  Over lap of the upper and lower incisors will be measured in millimeters.If incisors are missing, canines will be used.
Biofilm around the stainless steel crown as assessed by the Modified Plaque Index | 3 months post intervention
  In the Modified Plaque Index, a score of 0 (no plaque), 1 (thin visible plaque, difficult to identify), or 2 (thick visible plaque, easily detected) is assigned
Biofilm around the stainless steel crown as assessed by the Modified Plaque Index | 6 months post intervention
  In the Modified Plaque Index, a score of 0 (no plaque), 1 (thin visible plaque, difficult to identify), or 2 (thick visible plaque, easily detected) is assigned
Biofilm around the stainless steel crown as assessed by the Modified Plaque Index | 9 months post intervention
  In the Modified Plaque Index, a score of 0 (no plaque), 1 (thin visible plaque, difficult to identify), or 2 (thick visible plaque, easily detected) is assigned
Biofilm around the stainless steel crown as assessed by the Modified Plaque Index | 12 months post intervention
  In the Modified Plaque Index, a score of 0 (no plaque), 1 (thin visible plaque, difficult to identify), or 2 (thick visible plaque, easily detected) is assigned
Gingival health of the treated tooth as assessed by gingival status score | 3 months post intervention
  Gingival status is assigned a score of 0 (normal gingiva, natural coral pink gingival with no e/o inflammation), 1 (mild inflammation, slight changes in color, slight edema, no bleeding on probing), 2 (moderate inflammation, redness, edema, and glazing, bleeding on probing), or 3 (severe inflammation, marked redness and edema/ulceration/tendency to bleed spontaneously).
Gingival health of the treated tooth as assessed by gingival status score | 6 months post intervention
  Gingival status is assigned a score of 0 (normal gingiva, natural coral pink gingival with no e/o inflammation), 1 (mild inflammation, slight changes in color, slight edema, no bleeding on probing), 2 (moderate inflammation, redness, edema, and glazing, bleeding on probing), or 3 (severe inflammation, marked redness and edema/ulceration/tendency to bleed spontaneously).
Gingival health of the treated tooth as assessed by gingival status score | 9 months post intervention
  Gingival status is assigned a score of 0 (normal gingiva, natural coral pink gingival with no e/o inflammation), 1 (mild inflammation, slight changes in color, slight edema, no bleeding on probing), 2 (moderate inflammation, redness, edema, and glazing, bleeding on probing), or 3 (severe inflammation, marked redness and edema/ulceration/tendency to bleed spontaneously).
Gingival health of the treated tooth as assessed by gingival status score | 12 months post intervention
  Gingival status is assigned a score of 0 (normal gingiva, natural coral pink gingival with no e/o inflammation), 1 (mild inflammation, slight changes in color, slight edema, no bleeding on probing), 2 (moderate inflammation, redness, edema, and glazing, bleeding on probing), or 3 (severe inflammation, marked redness and edema/ulceration/tendency to bleed spontaneously).

CONTACTS AND LOCATIONS:
Overall Officials: Nathanael O Salako, BDS,MSc, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No